CLINICAL TRIAL: NCT03388866
Title: Effect of Sublingual Immunotherapy With Mite Extract in Patients With Atopic Dermatits: Placebo-controlled Double-blind Randomized Study
Brief Title: Effect of Sublingual Immunotherapy in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Casa Espirita Terra de Ismael (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Fabio Carmona, Head of Medical School of Ribeirão Preto - University of São Paulo Children´s Hospital, Casa Espirita Terra de Ismael
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SLIT_AD1
Record Dates: First submitted 2017-11-22; First posted 2018-01-03 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Atopic Dermatitis; Effects of Immunotherapy
Keywords: inhaled aeroallergens; eczema; pruritus; life quality; immunotheraphy; atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Intervention Model Description: A total of 94 patients, 3 years of age or older, with clinical diagnosis of AD, without distinction of gender, ethnicity or social group, will be selected at HCFMRP-USP Allergy and Dermatology outpatient clinics. These patients will undergo clinical evaluation and laboratory tests, including blood count, total IgE, inhalant panel specific IgE, and / or immediate hypersensitivity skin tests, and mite allergen specific IgG4 (Der p 1 and Der p 2), before of the study.
  Patients in the treatment group will undergo sublingual allergen-specific immunotherapy with weekly and weekly doses of extracts of Dermatophagoides pteronyssinus and Dermatophagoides farinae mites (60% and 40% respectively), according to the predetermined schedule. Patients in the control group will be submitted to the same administration schedule, but with allergen extract diluent (doubly distilled water solution and glycerin).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects will be randomly divided into blocks of random size 4 or 6 and stratified according to age (less than 12 years and greater / equal 12 years) and severity (SCORAD less than 50 and greater / equal 50)**, performed through the RedCap platform, available at FMRPUSP. This process will be performed by laboratory staff who will provide the extracts and the researchers will not have access to the lists of patients in each group. As for blinding, the bottles with extract and placebo will be provided by the already coded laboratory, and the team will only be responsible for the delivery and storage of the same.
  ** Initial SCORAD was not part of the stratification because it was part of the primary outcome variable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mite extract sublingual immunotherapy (Active Comparator): Use of mite extract sublingual immunotherapy (SLIT) with increasing weekly doses of extracts of mite Dermatophagoides pteronyssinus, as represented below:
  Weekly dose schedule Monday Wednesday Friday
  1. st week 1 drop 2 drops 4 drops
  2. nd week 6 drops 8 drops 8 drops
  Monthly Dilution Schedule Dilution of mite extract
  1st and 2nd weeks (1st month) 1: 1000000 v: v 3rd and 4th weeks (1st month) 1: 100000 v: v
  1st and 2nd weeks (2nd month)1: 10000 v: v 3rd and 4th weeks (2nd month) 1:1000 v: v
  1st and 2nd weeks (3rd month) 1: 100 v:v 3rd and 4th weeks (3rd month) 1:10 v:v 3rd to 18th month 1:10 v: v
  Interventions: Drug: Mite extract sublingual immunotherapy (SLIT)
- SLIT placebo (Placebo Comparator): Patients in the control group will be submitted to the same administration schedule, but with allergen extract diluent (doubly distilled water solution and glycerin), as described below:
  Weekly dose schedule Monday Wednesday Friday
  1. st week 1 drop 2 drops 4 drops
  2. nd week 6 drops 8 drops 8 drops
  Intervention: Placebo - Immunotherapy allergen diluent
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mite extract sublingual immunotherapy (SLIT) — Administration of increasing weekly doses of extracts of mites Dermatophagoides pteronyssinus in the treatment group.
  Other Names: Allergen specific sublingual immunotherapy; Sublingual immunotherapy (SLIT)
  Arms: Mite extract sublingual immunotherapy
Other: Placebo — Placebo group will be submitted to administration of increasing weekly doses, but with diluent of the allergenic extract (doubly distilled water solution and glycerin).
  Other Names: Diluent of the allergenic extract
  Arms: SLIT placebo

SUMMARY:
Atopic dermatitis (AD) is a chronic and recurrent inflammatory disease, prevalent between 1 and 20% in the world population, with a predominance of childhood, but which may be present in adult life. AD results from a complex interaction between genetic and environmental factors, with the presence of a defect in the skin barrier and deregulation of the immune response, culminating in an inflammatory response in the skin predominantly type 2. Disease control is based on restoring skin hydration, smoothing itching and controlling the process specific sensitizing agents such as inhalant allergens and foods that may pathogenesis of the disease. In selected patients who present IgE mediated response to inhalant allergens, allergen-specific immunotherapy can be effective. Classically, the subcutaneous route is the most used, however, sublingual immunotherapy (SLIT) has been used in increasing form. There are still few studies on the efficacy and safety of SLIT in atopic dermatitis. Therefore, the present study aims to to investigate the role of SLIT in the management of patients with AD allergic mites, through a randomized, double-blind and placebo-controlled study

DETAILED DESCRIPTION:
A total of 94 patients, 3 years of age or older, with clinical diagnosis of AD, without distinction of gender, ethnicity or social group, will be selected at HCFMRP-USP Allergy and Dermatology outpatient clinics. These patients will undergo clinical evaluation and laboratory tests, including blood count, total IgE, inhalant panel specific IgE, and immediate hypersensitivity skin tests, and mite allergen-specific IgG4 (Der p 1 and Der p 2), before of the study. To calculate the sample size, a response rate to the medication was defined as a 15 - point decrease in SCORAD (a score that includes lesion extent, intensity and subjective symptoms such as pruritus and sleep), which was determined through the experience of the service. It was estimated that 40% of the patients in the treatment group and 15% of the placebo group reached the proposed rate through a test with 80% power, and the need for 47 individuals in each group was defined.

Patients in the treatment group will undergo allergen-specific immunotherapy sublingually, with weekly doses of extracts of mites Dermatophagoides pteronyssinus and Dermatophagoides farinae (60% and 40% respectively), according to the scheme described in Tables 1 and 2. Patients in the control group will be submitted to the same administration schedule, but with the diluent of the allergenic extract (doubly distilled water solution and glycerin). Patients will be divided into groups according to randomization.

Subjects will be randomly divided into blocks of random size 4 or 6 and stratified according to age (less than 12 years and greater / equal 12 years), performed through the RedCap platform, available at FMRPUSP. This process will be performed by laboratory staff who will provide the extracts and the researchers will not have access to the lists of patients in each group. As for blinding, the bottles with extract and placebo will be provided by the already coded laboratory, and the team will only be responsible for the delivery and storage of the same.

Table 1 - Weekly dose schedule Monday Wednesday Friday

1. st week 1 drop 2 drops 4 drops
2. nd week 6 drops 8 drops 8 drops

Table 2 - Monthly Dilution Schedule Dilution of mite extract

1st and 2nd weeks (1st month) 1: 1000000 v: v 3rd and 4th weeks (1st month) 1: 100000 v: v

1st and 2nd weeks (2nd month)1: 10000 v: v 3rd and 4th weeks (2nd month) 1:1000 v: v

1st and 2nd weeks (3rd month) 1: 100 v:v 3rd and 4th weeks (3rd month) 1:10 v:v 3rd to 18th month 1:10 v: v

Individuals will be the outpatient clinics of the Allergy and Dermatology Service of the HCFMRP-USP. All medical records and clinical and dermatological examination will be recorded in medical records, as well as clinical evaluation by SCORAD , quality of life questionnaire and personal scale of symptoms, being evaluated at the beginning of treatment, after two, three, six, nine, twelve, fifteen and eighteen months of evolution.

Serum levels of IgG4 specific mite for Der p 1 and Der p 2 will be determined by ImmunoCAP and evaluated at the beginning and the end of treatment. Interleukins 4, 5, 9, 10 13, 17, TNFα, TGFβ and interferon-γ will be performed in plasma in the beginning, with 9 months of evolution and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD according to Hanifin and Rajka criteria;
* Age greater than or equal to 3 years;
* SCORAD equal to or greater than 15 points;
* Presence of skin tests and / or specific IgE positive for Dermatophagoides pteronyssinus and / or Dermatophagoides farinae;

Exclusion Criteria:

* Pregnancy or breastfeeding;

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Decrease in Severity Scoring of Atopic Dermatitis (SCORAD) | Measures at baseline and after 18 months
  The SCORAD is calculated using the extent of the injury, intensity and subjective symptoms, the formula used for the calculation is A / 5 + 7B / 2 + C (A - extent B - intensity C-subjective symptoms). The extent can vary from zero to 100, applying the nine rule also used in large burned patients. The intensity varies from zero to 18, divided into six items, including erythema, edema, excoriation, lichenification, and dryness. Subjective symptoms range from zero to 30 evaluated by means of analog pruritus scale and sleep.
  The SCORAD severity rating is:
  0-20 mild 20-40 moderate > 40 severe
  Based on our clinical experience, it was decided to consider as the main outcome a 15-point decrease in SCORAD,in any degree of severity, in 40% of subjects in the treatment group and 15% in the placebo group.

SECONDARY OUTCOMES:
EASI (Eczema Area and Severity Index) | 3, 6, 9, 12, 15 and 18 months
  EASI is based on the extension and severity of Atopic Dermatitis. To obtain EASI, the proportion of body areas are taken into consideration, with head being equivalent to 10%, trunk 30%, upper extremities 20% and lower extremities 40%. The percentage of involvement of these four regions is determined using a scale of 0 to 6. Clinical signs including erythema, infiltration and/or papulation, excoriation, and lichenification are evaluated each on a scale of 0 to 3.
  Final score is calculated using the formula below. Severity is classified as: 0 = clear; 0.1 - 1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe. Any reduction in the EASI score will be accepted as a positive outcome.
IGA (Investigator Global Assessment) | 3,6,9,12,15 and 18 months
  IGA consists of evaluation of the severity of Atopic Dermatitis considering the inflammatory signs of the disease (erythema, papulation and infiltration). IGA is calculated according to the following scale: clear; almost clear; mild disease; moderate disease; severe disease; and very severe disease.
  IGA score 0 or 1 after 18 months of treatment will be accepted as a positive outcome.
DLQI (Dermatology Life Quality Index) | 3, 6, 9, 12,15 and 18 months
  The DLQI is a questionnaire of 10 questions used to measure how much skin problems affect patient´s life in the past seven days.
  The scoring of each question is as follows:
  Very much, score of 3; A lot, score of 2; A little, score of 1; Not at all, score of 0; Not relevant, score of 0. Question 7, 'prevented work or studying', score of 3. The DLQI is calculated by summing the score for each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  How to interpret meaning of DLQI scores:
  0 - 1 no effect at all on patient's life; 2 - 5 small effect on patient's life; 6 - 10 moderate effect on patient's life; 11 - 20 very large effect on patient's life; 21 - 30 extremely large effect on patient's life.
  The decrease of 4 or more points in DLQI is a secondary outcome measure.
Analog Visual Scale of Symptoms | 3, 6, 9, 12,15 and 18 months
  The analog visual scale consists of three questions that can be answered using a scale of 0 to 10, as described below:
  How much your skin itched last week? How much your skin peeled last week? How atopic dermatitis interfered with last week's sleep? Any reduction in the analog visual scale will be accepted as a positive outcome
Pruritus scale | 3, 6, 9, 12, 15 and 18 months
  Patients will provide information on their perception of pruritus in their daily life. The evaluation is subjective, varying from absence of pruritus to severe pruritus.
  Any reduction in the Pruritus scale will be accepted as a positive outcome
IgG4 antibodies to mite allergens Der p 1, Der p 2 and Der p 10 | 0 and 18 months
  It has been consistently shown that both subcutaneous and sublingual immunotherapy increase levels of specific IgG4 antibodies. Therefore, we expect to find an increase in levels of IgG4 to mite allergens at the end of treatment. IgG4 specific to Der p 1, Der p 2 and Der p 10 can be measured by ImmunoCAP.
Specific IgE antibodies to purified allergens and to Staphylococcal allerg | 0 and 18 months
  IgE antibodies to a panel of purified allergens will be assessed by ImmunoCAP and ImmunoCAP-ISAC, including Dermatophagoides pteronyssinus allergens rDer p1, rDer p 2 e rDer p 10. In addition, levels of specific IgE to Staphylococcal enterotoxins, including enterotoxins A, B, C and TSST, will be determined in patients' sera before and after treatment. It is expected that levels of IgE antibodies to mite allergens and to Staphylococcal enterotoxins will be decreased at the end of treatment
Type 2 and regulatory cytokines | 0, 9 and 18 months
  Reduction in type 2 cytokine group (IL4, IL5, IL9 and IL13) Regulatory cytokines [Time Frame: 0, 9 and 18 months] Increase of regulatory cytokines (IL-10 and TGF-beta)

CONTACTS AND LOCATIONS:
Overall Officials: Karla L Arruda, PhD, Study Director — Faculdade de Medicina de Ribeirão Preto
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided